CLINICAL TRIAL: NCT04943120
Title: Clinical Evaluation of "Snow-Plow" Technique Versus Bulk Fill Technique in Restoration of Class II Cavities: Randomized Clinical Trial
Brief Title: Clinical Evaluation of "Snow-plow"Technique Versus Bulk Fill Technique in Restorations of Class II Cavities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Mohamed Ahmed Gomaa, Main Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422019484260
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Class II Dental Caries

STUDY DESIGN:
Intervention Model Description: 1:1
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Snow-Plow" technique (Experimental): In class II cavities, application of X-tra Base bulk fill flowable composite (VOCO) in 1 mm thickness without curing followed by X-tra Fill bulk fill packable composite (VOCO) to restore the proximal wall. Polymerization as one unit for 20 seconds.
  Interventions: Procedure: "Snow-plow" technique
- Bulk Fill technique (Active Comparator): In class II cavities, application of 4 mm increment of X-tra Fill bulk fill packable composite (VOCO) to restore the proximal wall. then the restoration id fully polymerized.
  Interventions: Procedure: Bulk fill technique

INTERVENTIONS:
Procedure: "Snow-plow" technique — In class II cavities, application of X-tra Base bulk fill flowable composite (VOCO) in 1 mm thickness without curing followed by X-tra Fill bulk fill packable composite (VOCO) to restore the proximal wall. Polymerization as one unit for 20 seconds.
  Arms: "Snow-Plow" technique
Procedure: Bulk fill technique — In class II cavities, application of 4 mm increment of X-tra Fill bulk fill packable composite (VOCO) to restore the proximal wall. then the restoration id fully polymerized.
  Arms: Bulk Fill technique

SUMMARY:
The aim of the study is to assess the performance of " snow-plow" technique as compared to Bulk Fill technique in restoration of class II cavities.

DETAILED DESCRIPTION:
1. With limited evidence-based information about the clinical performance of resin composite in class II cavities. it is beneficial to compare the newly introduced "snow-plow' technique using a randomized clinical trial to test the null hypothesis that this new technique has the same clinical performance.
2. The comparator will be the bulk fill technique as an alternative to the conventional layering technique. This is because it has shown lower polymerization shrinkage when comparing it to the conventional composite. Bulk fill has reduced the chair time for the patient. It is done by the application of 4mm increment and cured at once.
3. Patients are selected according to the eligibility criteria discussed in the following section.
4. local anesthesia will be administered and the operative field will be isolated before starting the restorative procedure. A standard class II cavity will be prepared at the two-surface cavities.
5. The preparation will be performed using rotary instrumentation for cavity preparation by a water-cooled high-speed hand-piece by the same operator.
6. The teeth are then restored using one of the two techniques according to their allocation with the same steps discussed in the different arms.
7. The restorations are assessed using the modified USPHS criteria at the time intervals stated in the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* class II carious lesions in premolars and molars.
* Vital upper or lower teeth with no signs of irreversible pulpitis.
* Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth.

Exclusion Criteria:

* Deep carious defects (close to pulp, less than 1 mm distance).
* Periapical pathology or signs of pulpal pathology.
* Endodontically treated teeth
* Tooth hypersensitivity.
* Possible prosthodontic restoration of teeth.
* Heavy occlusion or occlusal contacts or history of bruxism.
* Severe periodontal affection.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
clinical performance | day 1
  USPHS Criteria
clinical performance | 3 months
  USPHS Criteria
clinical performance | 6 months
  USPHS Criteria
clinical performance | 9 months
  USPHS Criteria
clinical performance | 12 months
  USPHS Criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No